CLINICAL TRIAL: NCT06062303
Title: Hemodynamic Phenotype-Based, Capillary Refill Time-Targeted Resuscitation In Early Septic Shock: The ANDROMEDA-SHOCK-2 Randomized Clinical Trial (A2)
Brief Title: Hemodynamic Phenotype-Based,Capillary Refill Time-Targeted Resuscitation In Early Septic Shock:ANDROMEDA-SHOCK-2
Acronym: ANDROMEDA-FR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP220794
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Intensive Care Unit Acquired Weakness; Shock, Septic
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: comparative multicentre, open-label, investigator-led randomized controlled trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compartor arm (No Intervention): - Patients allocated to the usual care group will be managed by the clinical staff according to usual practice at their sites including decisions about hemodynamic and perfusion monitoring, and all treatments, but should follow general recommendations of the Surviving Sepsis Campaign to avoid extremes of clinical practice. This includes basic hemodynamic targets such as a MAP >65 mmHg, HR (heart rate) <120 beats per minute (BPM), arterial oxygen saturation (SaO2) >94%, Hb > 7 gr/dl, and the use of NE as the first vasopressor and crystalloids as the fluid of choice.
- Capillary-refill time and phenotyping group (Active Comparator): Patients w/normal baseline CRT will be periodically monitored. Patients with abnormal CRT and septic shock will be categorized according to pulse pressure (PP). If <40 mmHg, will go to fluid responsiveness (FR) assessment. FR (-) patients will undergo cardiac echo to rule out significant dysfunction. Fluid boluses will be administered in 30 min intervals and repeated as needed if CRT is still abnormal. Patients with PP ≥40 mmHg will proceed according to diastolic pressure (DAP). If ≥50 mmHg will move to FR assessment. If <50 mmHg NE will be increased for MAP >65 mmHg and DAP ≥50 mmHg w/CRT assessed 1 h after. NE will be increased in 0.1 mcg/k/m increments up to 0.5 mcg/k/m.
  If CRT is normal, patients will proceed to periodic monitoring. Patients with persistent abnormal CRT or that reached NE safety limit will proceed directly to echo.
  Patients that correct CRT with first tier interventions will not be subjected to obligatory echo but will just proceed to periodic monitoring.
  Interventions: Other: Usual care (UC)

INTERVENTIONS:
Other: Usual care (UC) — - Patients allocated to the UC group will be managed by the clinical staff according to usual practice at their sites including decisions about hemodynamic and perfusion monitoring, and all treatments, but should follow general recommendations of the Surviving Sepsis Campaign to avoid extremes of clinical practice. This includes basic hemodynamic targets such as a MAP >65 mmHg, heart rate (HR) <120 beats per minute (BPM), arterial oxygen saturation (SaO2) >94%, Hb > 7 gr/dl, and the use of NE as the first vasopressor and crystalloids as the fluid of choice.
  Arms: Capillary-refill time and phenotyping group

SUMMARY:
Over-resuscitation including fluid overload has been associated with increased morbidity (prolonged duration of organ failure) and mortality in septic shock. "One-size-fits-all" resuscitation strategies may increase septic shock mortality. However, clinical studies on individualized resuscitation are lacking. Hemodynamic phenotyping may allow to individualize septic shock resuscitation. The ANDROMEDA-SHOCK trial found that a simple clinical and bedside CRT-targeted resuscitation reduces organ dysfunction and 28-day mortality in septic shock. The current study will examine the hypothesis that a CRT-targeted resuscitation based on hemodynamic phenotyping considering within an decision tree usual bedside clinical parameters such as pulse pressure, diastolic blood pressure, fluid responsiveness and cardiac performance can further decrease mortality in septic shock as compared to usual care.

DETAILED DESCRIPTION:
Septic shock is associated with a high mortality risk related to progressive tissue hypoperfusion.However, despite extensive research on the best monitoring and resuscitation strategies, many uncertainties remain. Over-resuscitation, particularly when inducing fluid overload, might contribute to a worse outcome. Fluid overload more likely occurs when fluids are administered to fluid unresponsive patients, but also when inappropriate resuscitation goals are pursued, or a "one-size-fit all" strategy is followed. From a hemodynamic point of view, several pathogenic mechanisms determine a progressive circulatory dysfunction While loss of vascular tone and relative hypovolemia predominate in early phases, more complex mechanisms such as endothelial and microcirculatory dysfunction, progressive vasoplegia, and myocardial dysfunction may be involved later. In effect, from a clinical point of view, many patients despite been fluid loaded in pre-intensive care unit settings, are still evidently hypovolemic and benefit from further administration of fluid boluses. Others, however, present very low diastolic arterial pressures reflecting profound vasoplegia, and recent data suggest that these patients may benefit from early norepinephrine instead of fluids[; on the contrary, administering fluids may fail to correct vascular tone and increase the risk of fluid overload[2]. In addition, a recent echocardiography-based study confirms that a relevant myocardial dysfunction is present in a significant number of patients, and that several cardiovascular phenotypes with a potentially different therapeutic approach may be recognized[8]. Unfortunately, despite the availability of most of the parameters at the bedside and research efforts, no universally applicable clinical phenotyping method for septic shock patients has been translated to usual practice. This is particularly problematic since chocardiography is not immediately available in the majority of centers worldwide, and therefore initial decisions on fluid resuscitation are usually based on clinical grounds and tend to follow the one-size-fits-all principle, leading to the risk of fluid overload.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients (≥ 18 years)
* Patients with septic shock according to Sepsis-3 consensus conference. In short, septic shock is defined as suspected or confirmed infection, plus hyperlactatemia and NE requirements due to persistent hypotension, after a fluid load of at least 1000mL in 1h
* Patient and/or relative informed and having signed the information and consent form for participation in the study

Exclusion Criteria:

* More than 4 hours since septic shock diagnosis,
* Anticipated surgery or acute hemodialysis procedure to start during the 6h intervention period
* Active bleeding,
* Do not resuscitate status,
* Child B-C Cirrhosis
* Underlying disease process with a life expectancy < 90 days and/or the attending clinician deems aggressive resuscitation unsuitable
* Refractory shock (high risk of death within 24h)
* Pregnancy
* Concomitant severe acute respiratory distress syndrome
* Patients in whom CRT cannot be accurately assessed
* Non-affiliation to a social security scheme or to another social protection scheme
* Patient on AME (state medical aid) (unless exemption from affiliation
* Patient under legal protection (guardianship, curatorship)
* Participation in another interventional study involving human participants or being in the exclusion period at the end of a previous study involving human participants, if applicable
* Inability, according to the investigator, to understand the study (non-French-speaking patient, cognitive disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
A composite of all cause 28-days mortality plus time to cessation of vital support and length of hospital stay | 28 days
  A hierarchical composite of all cause mortality within 28 days, time to cessation of vital support (truncated at 28 days) and length of hospital stay (truncated at 28 days).

SECONDARY OUTCOMES:
All-cause mortality within 28 days | 28 days
  All-cause mortality within 28 days
Vital support free days | 28 days
  The number of calendar days between randomization and 28 days that the patient is alive and with no requirement of cardiovascular, respiratory and renal support. Patients who die within 28 days will have zero days counted for this variable, irrespective of vital support status.
  Resolution of cardiovascular failure implies complete stopping of vasopressor support for at least 24 consecutive hours. Resolution of respiratory failure implies extubation / liberation from mechanical ventilation for at least 48 hours. Resolution of renal failure implies liberation of renal replacement therapy for at least 72 hours in those receiving continuous replacement modalities and at least 5 days for those receiving intermittent ones.
Length of hospital stay | 28 days
  Number of days remaining hospitalized (from randomization up to hospital discharge), truncated at day 28.

OTHER OUTCOMES:
Length of ICU stay | 28 days
  Number of days remaining in ICU (from randomization up to ICU discharge). Re-admission to ICU during follow-up period will be accounted for the original ICU length of stay only if occurred within the next week of ICU discharge and by a cause related with the original admission.
Time to cessation of vasopressor support | 28 days
  The number of hours between randomization and complete stopping of vasopressor support (defined as its complete interruption for at least 24 consecutive hours), within 28 days from randomization
Time to cessation of mechanical ventilation | 28 days
  The number of calendar days between intubation / start of mechanical ventilation and extubation / liberation from mechanical ventilation (maintained for at least 48 hours) within 28 days from randomization.
Time to cessation of renal replacement therapy | 28 days
  The number of calendar days between start of renal replacement therapy and complete liberation from renal replacement therapy (at least 48 hours for continuous replacement modalities and 5 days for intermittent ones) within 28 days from randomization.
Vasopressor support-free days | 28 days
  The number of calendar days without vasopressor support from randomization up to day 28. Cessation of vasopressor support implies its complete interruption for at least 24 consecutive hours.
Mechanical ventilation-free days | 28 days
  The number of calendar days without mechanical ventilation support from randomization up to day 28. Cessation of mechanical ventilation support implies its complete interruption for at least 48 consecutive hours.
  Re-start of mechanical ventilation during follow-up period will be accounted for the original mechanical ventilation-free days only if this occurs within the next week of ICU discharge and by a cause related with the original admission.
Renal replacement therapy-free days | 28 days
  The number of calendar days without renal replacement therapy from randomization up to day 28. Cessation of renal replacement therapy implies its complete interruption for at least 72 hours in those receiving continuous replacement modalities and at least 5 days for those receiving intermittent ones.
  Re-start of renal replacement therapy during follow-up period will be accounted for the original renal replacement-free days only if this occurs within the next week of ICU discharge and by a cause related with the original admission.
Variation in Sequential Organ Failure Assessment (SOFA) score | 7 days
  The Sequential Organ Failure Assessment (SOFA) is used to track a patient's status during the stay in the ICU to determine the extent of organ dysfunction. Its values ranges from 0 to 24. Higher SOFA scores associate with a worse outcome.
  The SOFA score will be calculated upon the maximum values observed on the day of enrollment and then, at days 2, 3, 4, 5 and 7 (or until patient discharge or death, if this happened before day-7), using clinically available data. If an individual organ dysfunction value is not available (i.e., cardiovascular, respiratory, renal, etc.), it will be assumed to be zero unless previous value was abnormal (in which case it would be considered the same organ score). Neurological score under sedation/invasive mechanical ventilation will be computed as that observed just before sedation/intubation.
Variation of creatinine-based KDIGO stage | 7 days
  Renal function assessed according to "Kidney Disease: Improving Global Outcomes (KDIGO) staging system from randomization through day 7 to assess for "de novo" or "worsening" acute kidney injury. Patients under chronic renal replacement therapy will not meet this end-point
Volume of resuscitation fluids | 72 hours
  The volume of fluids administered with resuscitative intention up to 72 hours from randomization.
Net fluid balance | 72 hours
  The volume of cumulated fluids during the first 72 hours from randomization.
Evolvement of capillary refill time (CRT) | 72 hours
  Evolvement of CRT within the first 72 hours after randomization.
Evolvement of lactate levels | 72 hours
  Evolvement of arterial lactate levels within the first 72 hours after randomization.
Evolvement of central venous pressure | 72 hours
  Evolvement of Central venous pressure within the first 72 hours after randomization.
Evolvement of central venous oxygen saturation | 72 hours
  Evolvement of central venous oxygen saturation within the first 72 hours after randomization
Evolvement of central venous to arterial carbon dioxide difference | 72 hours
  Evolvement of central venous to arterial carbon dioxide difference within the first 72 hours after randomization.
All-cause mortality within 90 days | 90 days
  All-cause mortality within 90 days
Length of hospital stay | 90 days
  Number of days remaining hospitalized (from randomization up to hospital discharge), truncated at day 90.
Changes in CRT before and after fluid resuscitation or increase in norepinephrine | 72 hours
  Assess the changes in CRT before and after fluid resuscitation or increase in norepinephrine doses and analyse their correlation with changes in haemodynamic parameters: systolic arterial pressure (SAP), diastolic arterial pressure (DAP), mean arterial pressure (MAP), pulse pressure (PP), cardiac output (CO) when available.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Robert Debré, Université de Reims, Reims, France